CLINICAL TRIAL: NCT00641836
Title: One-Year Follow-Up of Autologous Endothelial Progenitor Cells Transplantation in Patients With Idiopathic Pulmonary Arterial Hypertension
Brief Title: Safety and Feasibility of Autologous Endothelial Progenitor Cells Transplantation in Patients With Idiopathic Pulmonary Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPAH-EPC-2
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Idiopathic Pulmonary Arterial Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

INTERVENTIONS:
Procedure: Transplantation of autologous endothelial progenitor cells

SUMMARY:
Recent researches indicate that impairment of vascular and endothelial homeostasis plays a major role in the initiation and development of IPAH.We have recently reported the safety and feasibility data for autologous endothelial progenitor cells (EPCs) injection in patients with IPAH. Yet many questions remain unanswered: what is the ideal quantity of EPCs for therapy, the duration of the therapeutic effect, and moreover, the potential toxicity of such therapy. To help answer these questions, we designed the one year follow-up to investigate the safety and efficacy of autologous EPCs injection in patients with IPAH.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria included a base-line six minute walking distance between 100 and 450 m
* A resting mean pulmonary-artery pressure greater than 30 mm Hg
* A pulmonarycapillary wedge pressure of less than 15 mm Hg
* Pulmonary vascular resistance greater than 240 dyn•sec•cm-5
* 18-60 years old

Exclusion Criteria:

* The exclusion criteria included secondary pulmonary hypertension as a result of heart disease
* Pulmonary disease
* Sleep-associated disorders
* Chronic thromboembolic disease
* Autoimmune or collagen vascular disease
* HIV infection
* Liver disease
* New York Heart Association functional class IV
* Major bleeding requiring blood transfusion
* Diabetes
* Renal dysfunction
* Evidence for malignant diseases were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2005-07; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junzhu Chen, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- Department of Cardiology, the First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Result] Wang XX, Zhang FR, Shang YP, Zhu JH, Xie XD, Tao QM, Zhu JH, Chen JZ. Transplantation of autologous endothelial progenitor cells may be beneficial in patients with idiopathic pulmonary arterial hypertension: a pilot randomized controlled trial. J Am Coll Cardiol. 2007 Apr 10;49(14):1566-71. doi: 10.1016/j.jacc.2006.12.037. Epub 2007 Mar 27. PMID 17418297